CLINICAL TRIAL: NCT00372762
Title: Bumetanide Has a More Favourable Effect on Insulin Resistance Than Furosemide in Patients With Heart Failure - A Pilot Study
Brief Title: Bumetanide Versus Furosemide in Heart Failure
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to changes within the research program this study is not feasible at this time
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Neville Suskin, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-06-415
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Heart Failure
Keywords: Insulin resistance; heart failure; diuretic therapy
MeSH Terms: conditions — Heart Failure; Insulin Resistance | interventions — Furosemide; Bumetanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide (Active Comparator): Patients will be assigned to furosemide therapy (20mg to 80mg) orally, once or twice daily for an 8-week period.
  Interventions: Drug: Furosemide
- Bumetanide (Active Comparator): Patients will be assigned to bumetanide therapy at an equipotent dose to furosemide therapy (1mg bumetanide is equivalent to 40mg furosemide)for an 8-week period.
  Interventions: Drug: Bumetanide

INTERVENTIONS:
Drug: Furosemide — Current dose of furosemide will be maintained and equivalent dose bumetanide will be used following crossover
  Other Names: Lasix
  Arms: Furosemide
Drug: Bumetanide — Equivalent dose to pre-existing furosemide will be used
  Other Names: Bumex; Burinex
  Arms: Bumetanide
Drug: furosemide — 20mg to 80mg orally once or twice daily
  Other Names: Lasix
  Arms: Furosemide
Drug: bumetanide — 0.5mg to 2mg orally once or twice daily
  Other Names: Bumex; Burinex
  Arms: Bumetanide

SUMMARY:
Patients with NYHA FC II-III heart failure will be randomized in a cross-over fashion to 8 weeks of bumetanide versus furosemide therapy (equipotent dose), to test whether bumetanide therapy has a superior effect on insulin resistance compared to furosemide. Patients will be subject to a frequently sampled intravenous glucose tolerance test (FSIGT) with minimal model (MINMOD) analysis to assess insulin resistance and to a 6-minute walk test (6MWT) to assess functional capacity; patient recruitment and retention success, as well as medication adherence, will also be assessed.

DETAILED DESCRIPTION:
Insulin resistance is common in patients with heart failure (HF) and is associated with a worse functional capacity and more severe symptoms of heart failure. The majority of HF patients take furosemide on at least a daily basis for symptom relief. Bumetanide is a loop diuretic with a similar therapeutic diuretic effect to furosemide. There is evidence from observational and small comparative trials that bumetanide has a significantly less deleterious effect on indirect measures of insulin resistance compared with furosemide. However, a formal comparison between the 2 drugs using rigorous measures of insulin resistance has never been conducted in patients with HF. If bumetanide can be demonstrated to have a similar diuretic and a superior (less deleterious) effect on insulin resistance in patients with HF, the potential exists for bumetanide to have a significantly reduced morbidity in patients with heart failure compared to furosemide. In order to prepare for such a study, the variance of the MINMOD-derived insulin resistance from the FSIGT (26), in this group of patient needs to be determined along with the feasibility of conducting such a study. Functional capacity will be determined by duplicate 6-minute walk tests.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years of age
2. NHYA FC II or III HF AND documented LVEF ≤40% within 6 months prior to study entry
3. Taking 20 mg to 80 mg furosemide orally once or twice per day
4. No changes to cardiac medications for 3 months prior to study entry and no anticipated changes of medications for the duration of the study
5. No changes to oral anti-diabetic medications (if applicable) for 3 months prior to study entry, and no anticipated changes for the duration of the study (metformin, sulphonylurea type, glitazone type)
6. Ability to provide written consent

Exclusion Criteria:

1. Known sensitivity to bumetanide
2. Myocardial infarction, coronary angioplasty, coronary artery bypass surgery, admission for HF or unstable angina within a 3 month period prior to study recruitment
3. Planned coronary intervention within 6 months
4. Patients who are taking insulin
5. Patients with chronic renal (serum creatinine ≥ 200 μmol/L) or hepatic impairment (known cirrhosis or AST or ALT > 1.5 x upper limit of normal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance, as determined by frequently sampled intravenous glucose tolerance test with minimal model analysis (FSIGT MINMOD) | 3 months

SECONDARY OUTCOMES:
Fasting blood glucose | 3 months
Glycosylated hemoglobin (HbA1c) | 3 months
Serum creatinine, sodium, potassium, and chloride | 3 months
Submaximal exercise capacity as determined by the 6-minute walk test | 3 months
New York Heart Association Function Class heart failure (NYHA FC) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Neville G Suskin, MBChB, MSc, Principal Investigator — LHSC, University of Western Ontario
Locations (1):
- University Hospital, London Health Sciences Centre, London, Ontario, Canada